CLINICAL TRIAL: NCT06912191
Title: Investigating How the RECT Impacts Brain Functional States Through the ACC-cerebellar Loop
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Liqing Yao, Director, Department of Rehabilitation Medicine, the Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shen-PJ-Ke-2024-138
Record Dates: First submitted 2025-03-29; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Post-stroke Depression
Keywords: EEG; ERP

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- LC TMS combined with the RECT task (Experiment1) (Experimental): Left cerebellar single-pulse TMS stimulation combined with the RECT task
  Interventions: Other: Left cerebellar TMS stimulation combined with the RECT task
- RC TMS combined with the RECT task (Experiment1) (Experimental): Right cerebellar single-pulse TMS stimulation combined with the RECT task
  Interventions: Other: Right cerebellar TMS stimulation combined with the RECT task
- MC TMS combined with the RECT task (Experiment1) (Experimental): Midline cerebellar single-pulse TMS stimulation combined with the RECT task
  Interventions: Other: Midline cerebellar TMS stimulation combined with the RECT task
- Sham cerebellar single-pulse TMS stimulation combined with the RECT task (Experiment1) (Sham Comparator): Sham cerebellar single-pulse TMS stimulation combined with the RECT task, The TMS coil was placed at the cerebellar site but tilted 90° to prevent effective magnetic field penetration.
  Interventions: Other: Sham cerebellar TMS stimulation combined with the RECT task
- Combined Stimulus Intervention group （Experiment 2） (Experimental): Combined iTBS stimulation of the dorsolateral prefrontal cortex and TMS of the cerebellum with the RECT task intervention group
  Interventions: Other: The best stimulation protocol combined with left dorsolateral prefrontal cortex iTBS
- iTBS treatment group（Experiment 2） (Experimental): The group of participants will receive left dorsolateral prefrontal cortex iTBS stimulation, as well as sham cerebellar TMS stimulation and sham RECT task.
  Interventions: Other: Left dorsolateral prefrontal cortex iTBS stimulation, as well as sham TMS stimulation and sham RECT task.
- Traditional treatment group（Experiment 2） (Sham Comparator): The group of participants will receive sham left dorsolateral prefrontal cortex iTBS stimulation, sham cerebellar TMS stimulation, and sham RECT task.
  Interventions: Other: Sham left dorsolateral prefrontal cortex iTBS stimulation, sham cerebellar TMS stimulation, and sham RECT task.

INTERVENTIONS:
Other: Left cerebellar TMS stimulation combined with the RECT task — The first group will receive left cerebellar single-pulse TMS stimulation combined with the RECT task. RECT refers to rostral anterior cingulate cortexr (rACC)-engaging cognitive task. The theoretical basis of this task is that when subjects are in a state of focused attention, the power of theta neural oscillations in the midline of their frontal lobe will increase. By considering the features of post-stroke depression, this study combines the emotional recognition task with the RECT task. During each trial, individuals will view 4 faces consecutively, each displaying a different expression, and they will be required to memorize the sequence of expressions. Emoticons consist of joy, sorrow, and rage. After displaying four facial expressions, a brief text flowchart will appear. Participants need to check if the sequence reflected in the flowchart matches the order in which the four facial expressions appeared. If they match, click the left mouse button; if they do not match, click the
  Other Names: RECT task; TMS
  Arms: LC TMS combined with the RECT task (Experiment1)
Other: Right cerebellar TMS stimulation combined with the RECT task — Right cerebellar single-pulse TMS stimulation combined with the RECT task
  Other Names: RECT task; TMS
  Arms: RC TMS combined with the RECT task (Experiment1)
Other: Midline cerebellar TMS stimulation combined with the RECT task — Midline cerebellar single-pulse TMS stimulation combined with the RECT task
  Other Names: RECT task; TMS
  Arms: MC TMS combined with the RECT task (Experiment1)
Other: Sham cerebellar TMS stimulation combined with the RECT task — Sham cerebellar single-pulse TMS stimulation combined with the RECT task, The TMS coil was placed at the cerebellar site but tilted 90° to prevent effective magnetic field penetration.
  Other Names: RECT task
  Arms: Sham cerebellar single-pulse TMS stimulation combined with the RECT task (Experiment1)
Other: The best stimulation protocol combined with left dorsolateral prefrontal cortex iTBS — The optimal stimulation protocol determined in Experiment 1 combined with stimulation of the left dorsolateral prefrontal cortex.
  Other Names: left dorsolateral prefrontal cortex iTBS; RECT task; TMS
  Arms: Combined Stimulus Intervention group （Experiment 2）
Other: Left dorsolateral prefrontal cortex iTBS stimulation, as well as sham TMS stimulation and sham RECT task. — Subjects in the group underwent left dorsolateral prefrontal cortex iTBS stimulation, in addition to receiving sham TMS stimulation and participating in a sham RECT task. The sham RECT task involves having participants watch a continuous scroll of faces without needing to react.
  Other Names: left dorsolateral prefrontal cortex iTBS
  Arms: iTBS treatment group（Experiment 2）
Other: Sham left dorsolateral prefrontal cortex iTBS stimulation, sham cerebellar TMS stimulation, and sham RECT task. — The participants in this group received sham left dorsolateral prefrontal cortex iTBS stimulation, sham cerebellar TMS stimulation, and sham RECT task.
  Arms: Traditional treatment group（Experiment 2）

SUMMARY:
Experiment1: Using a brain EEG-TMS combined system, researchers aim to investigate the impact of the rostral anterior cingulate cortexr (rACC)-engaging cognitive task (RECT) combined single-pulse TMS magnetic stimulation on theta neural oscillations in the medial frontal lobe. The study will be divided into 4 groups: the first group will receive left cerebellar single-pulse TMS stimulation combined with the RECT task, the second group will receive right cerebellar single-pulse TMS stimulation combined with the RECT task, the third group will receive midline cerebellar single-pulse TMS stimulation combined with the RECT task, and the fourth group will receive sham cerebellar single-pulse TMS stimulation combined with the RECT task. Divide the participants into groups of 15 people each, following a 1:1:1:1 ratio. Based on the above testing, the stimulus method that results in the most significant change in the midline of the frontal lobe will be identified.

Experiment 2: Based on the research from Experiment 1, the most significant approach affecting theta neural oscillations in the medial frontal gyrus will be identified. This stimulation protocol will be combined with left dorsolateral prefrontal cortex iTBS stimulation in Experiment 2. The research aim of Experiment 2 is to investigate the most effective stimulation method for enhancing midline theta neural oscillations in the frontal lobe, in combination with left dorsolateral prefrontal cortex iTBS, for the treatment of post-stroke depression patients. This study will include 40 post-stroke depressed patients, and each participant must meet the inclusion criteria. The first group of participants, consisting of 20 individuals, will receive the optimal combination intervention. The second group of participants will only receive iTBS stimulation, without any additional intervention strategies used in Experiment 1. Patients will undergo Hamilton Depression Scale assessment and resting state and task state EEG collection at baseline, one week after intervention, and two weeks after intervention.The primary outcome will be the Hamilton Depression Scale, with EEG-related data being analyzed as a secondary outcome. Task-oriented EEG detection will include both facial expression recognition paradigm and oddball experiment paradigm. Reaction time, accuracy, and completion status will be recorded simultaneously in the experiment. The experiment will record patients' tolerance and any adverse events that occur.

ELIGIBILITY:
Inclusion Criteria:

* Onset of stroke <6 months ago, or >6 months since the last stroke event;
* Age >=18 years and <85 years (as the probability of Vascular Cognitive Impairment increases above 85);
* Patients with damage in the middle cerebral artery territory;
* NIHSS >4 and <26;
* mRS score >=2;
* Completion of CT or MRI;
* No neurological or psychiatric disorders; no impairment of consciousness; able to comply with relevant treatments; no severe cognitive dysfunction (MMSE >=15);
* All participants are right-handed; Sign the informed consent form.

Exclusion Criteria:

* History of epilepsy or psychiatric disorders (including depression, anxiety, or schizophrenia);
* Severe comorbidities;
* History of medication use: benzodiazepines, baclofen, antidepressants;
* Non-compliance with the treatment plan;
* Acute-phase cerebral hemorrhage, acute infectious diseases;
* Severe suicidal tendencies in individuals with depression;
* Individuals suffering from severe headaches, high blood pressure, malignant tumors, open wounds, vascular embolism, leukopenia, etc.;
* Severe alcohol abuse;
* History of cranial surgery, individuals with metal implants in the brain;
* Individuals with an implanted cardiac pacemaker;
* NIHSS >26, MMSE <15;
* Any disease likely to prevent the patient from surviving more than one month;
* Pregnant individuals.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale，MADRS | Day1
  This scale will be the primary outcome measure for Experiment 2. Montgomery-Asberg Depression Rating Scale，MADRS: Extreme depression: MADRS >35; Major depression: MADRS >30; Moderate depression: MADRS >22; Mild depression: MADRS >12; Remission stage: MADRS <12.
Electroencephalogram | Day 1
  EEG will be the main outcome measures for Experiment 1 and Experiment 2. EEG power in the delta, theta, alpha, beta band: the power spectral density (PSD) in unit^2/Hz Functional connectivity---Phase locking value (PLV): The value of PLV ranges from 0 to 1 Event related potentials in amplitude/μV

SECONDARY OUTCOMES:
Mini-mental state examination,MMSE | Day 1
  Mini-mental state examination,MMSE: A score of 27-30: normal; Score < 27: cognitive impairment.
Montreal Cognitive Assessment, MoCA | Day 1
  Montreal Cognitive Assessment, MoCA: The total score of the scale is 30 points, and the test result shows that the normal value is ≥26 points.
Hamilton Depression Scale，HAMD | Day 1
  Hamilton Depression Scale，HAMD: A total score of more than 35 May indicate severe depression.
Hamilton Anxiety Scale，HAMA | Day 1
  Hamilton Anxiety Scale，HAMA: The total score ≥29, may be severe anxiety; ≥21 points, there must be obvious anxiety; ≥14 points, definitely have anxiety; More than 7 points, may have anxiety; If the score is less than 7, there is no anxiety symptom
Quick Inventory of Depressive Symptomatology Self-Report, QIDS-SR16 | Day 1
  Quick Inventory of Depressive Symptomatology Self-Report, QIDS-SR16: The total score is calculated on a scale of 0 to 27, with higher scores being associated with higher levels of depression.
Response time | Day 1
  Recording their response times in seconds: The average reaction time of subjects in the facial expression recognition task to judge each facial expression picture.
Accuracy rates | Day 1
  Recording their accuracy rates in % during the task: The average correct rate at which subjects judged each expression picture in the facial expression recognition task.

IPD SHARING:
Plan to Share IPD: No